CLINICAL TRIAL: NCT06087666
Title: Integrating Families at Neonatal Intensive Care Units for Empowering Them as Primary Caregivres: the Impact of the Program
Brief Title: Alliance for Family Integrated Care Implementation in Neonatal Intensive Care Units
Acronym: RISEinFAMILY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 101007922
Record Dates: First submitted 2023-05-26; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Preterm
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: stepped wedge cluster controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FICare intervention (Experimental): FICare implementation model will be demonstrated by setting 5 pilots in non-FICare-experienced NICUs from NL, TR, RO, UK, ZM (AMC, GU, CLUJ, UHS, and UNZA, partners, respectively) and 2 pilots in clinical sites who have recently implemented FICare from ES and NL (SERMAS and OLVG).
  Interventions: Procedure: FICare
- control intervention (No Intervention): A cohort of patients born at the non-FICare clinical sites (AMC, GU, CLUJ, UHS, and UNZA) from the start of the study (November 2022) to the time assigned to start the intervention. A 3-month washout period will be established for staff training and site readiness.

INTERVENTIONS:
Procedure: FICare — The Family Integrated Care (FICare) programme has been developed in a multicenter cluster randomised controlled trial, with 26 tertiary NICUs from Canada, Australia and New Zealand, comparing standard NICU care (which was mainly care by nurses) (891 infants) to FICare programme (895 infants). FICare model and showed that the involvement of parents in the direct care improved weight gain and increased breastfeeding rates in the preterm infants. In addition, their parents had lower rates of stress and anxiety. These results were confirmed in a cluster-randomised controlled trial. Subsequent studies carried out so far have shown promising positive effects on a variety of domains. Maturation profiles have been shown to accelerate with the FICare intervention as a shorter time to achieve exclusive enteral nutrition as well as oral nutrition has been shown in the preterm infants included in FICARE programmes compared to control babies
  Arms: FICare intervention

SUMMARY:
International, multi-centre, pluri-cultural, stepped wedge cluster controlled trial, to demonstrate superiority of site tailored 'Family integrated care model'(FICare), that promotes the active participation of the parents as primary caregivers of their infants in neonatal intensive care units (NICU), versus standard NICU care delivery with regards to short-term health outcomes in high-risk newborns with prolonged hospital stay.

ELIGIBILITY:
Inclusion Criteria For infants :

1. Birth weight at or below 1500 g or gestational age at or below 34 weeks.
2. Any other peri-neonatal condition anticipating NICU specialised care.
3. Admission for at least 7 days
4. Decision to provide full life support.

Inclusion Criteria For Adults

1. Willingness to spend at least 6h per day at NICU OR commitment to attend educational sessions
2. Active involvement in care for their infant at least a 7 day-period
3. No intellectual or language barriers[A] to understanding
4. At least one primary caregivers involved in training [B]
5. Signed informed consent

Exclusion Criteria For Children:

1. Decision not to provide full life support
2. Critical illness unlikely to survive
3. Scheduled for early transfer to another non-FICare hospital (expected hospital stay <7days)

Exclusion Criteria for Parents:

1. Intellectual handicaps that makes difficult learning-understanding
2. Communication cannot be established even with translator
3. Mental, psychiatric problems or under legal supervision
4. Newborn under guardianship of social services
5. Lack of parental signed informed consent

Ages: 0 Weeks to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
RISEinFAMILY implementation: | Through study completion (average of 24 months)
  proportion of families completing basic and advanced training levels (observed vs expected).
RISEinFAMILY implementation: | Through study completion (average of 24 months)
  Average time to complete basic and advanced training levels (observed vs expected)
RISEinFAMILY implementation: | Through study completion (average of 24 months)
  Average time of kangaroo care per day
Short-term health infant's outcomes | Through study completion (average of 24 months)
  proportion of high-risk infants achieving and maintaining adequate growth patterns during NICU admission.

SECONDARY OUTCOMES:
Reported adverse event rate per 1000 patients/day | Through study completion (average of 24 months)
Feeding patterns at discharge: | Through study completion (average of 24 months)
  proportion of infants on exclusive breastfeeding
Brestfeeding rates at discharge: | Through study completion (average of 24 months)
  Number of patients with no breastfeeding
Brestfeeding rates at discharge: | Through study completion (average of 24 months)
  Number of patients with <50% of intake
Brestfeeding rates at discharge: | Through study completion (average of 24 months)
  Number of patients with >50% of intake
Parental psychological health | Through study completion (average of 24 months)
  Parental stress will be measured using the abbreviated Pediatric Stress Scale for Pediatric Intensive Care Unit (PSS PICU).
  Scale ranges from 0 to 5, higher scores indicate worse outcomes
Parental psychological health | Through study completion (average of 24 months)
  Anxiety and depression symptoms will be measured using the Four Item Patient health (PHQ-4).
  Scale ranges from 0 to 3, higher scores indicate worse outcomes
Parental psychological health | Through study completion (average of 24 months)
  Postnatal depression will be measured using the Edinburgh Postnatal Depression Scale (EPDS).
  Scale ranges from 0 to 3, higher scores indicate worse outcome.
Parental psychological health | Through study completion (average of 24 months)
  Maternal self-efficacy will be measured using the Perceived Maternal Parenting Self-Efficacy (PMP S-E).
  Scale ranges from 0 to 3, higher scores indicate better outcome
Parental psychological health | Through study completion (average of 24 months)
  Maternal-to-infant-bonding scale will be measured using the Maternal-to-Infant Bonding Scale.
  Score ranges 0 to 3. For items 1,2 and 6, higher scores correlate to better outcomes; for items 2, 3, 5, 7 and 8, higher scores correlate to a worse outcome.
Parental psychological health | Through study completion (average of 24 months)
  Resilience will be measured Brief Resilience Scale. Scale ranges from 0 yo 6. For items 4, 7, 9, 12, 17, 18, 19 and 21, higher scores indicate a better outcome. For items 1, 2, 3, 5, 6, 8, 10, 11, 13, 14, 15, 16m 20 and 22 a higher score indicates a worse outcome.
Feeding patterns at discharge: | Through study completion (average of 24 months)
  Day of life (DOL) to complete oral feeding (nasogastric tube removed)
Feeding patterns at discharge: | Through study completion (average of 24 months)
  day of life (DOL) to reach full enteral nutrition (>130 mL/K/day)
Feeding patterns at discharge: | Through study completion (average of 24 months)
  DOL at discharge
Proportion of infants diagnosed of (at 36 weeks PMA or discharge): bronchopulmonary dysplasia, oxygen dependency, severe retinopathy of prematurity (grade 3 or need for treatment), nosocomial infection necrotising enterocoli | Through study completion (average of 24 months)
Satisfaction and self-care of professionals measured by surveys | Through study completion (average of 24 months)
  Anxiety and depression symptoms will be measured using the anxiety and depression survey (PHQ-4).
  The scale ranges from 1 to 3. Higher scores indicate a worse outcome.
Satisfaction and self-care of professionals measured by surveys | Through study completion (average of 24 months)
  burnout symptoms will be measured using the Maslach burnout inventory human services survey (MBI-HSS). Scale ranges from 0 to 6. For Items 4, 7, 9, 12, 17, 18, 19 and 21, higher scores indicate a better outcome. For items 1, 2, 3, 5, 6, 8, 10, 11, 13, 14, 15, 16, 20 and 22, higher scores indicate a worse outcome.
Satisfaction and self-care of professionals measured by surveys | Through study completion (average of 24 months)
  post-traumatic stress will be measured using (post traumatic stress survey (PTSD-8). Scale ranges from 0 to 3, higher scores indicate worse outcomes
Satisfaction and self-care of professionals measured by surveys | Through study completion (average of 24 months)
  Work and wellbeing will be measured using Unwes-9 work and well-being survey (UWES).
  Scale ranges from 0 to 6, a higher score indicates a better outcome
Feeding patterns at discharge: | Through study completion (average of 24 months)
  postmenstrual age (PMA) to complete oral feeding (nasogastric tube removed)
Feeding patterns at discharge: | Through study completion (average of 24 months)
  postmenstrual age (PMA) to reach full enteral nutrition (>130 mL/K/day)
Feeding patterns at discharge: | Through study completion (average of 24 months)
  postmenstrual age (PMA) at discharge

OTHER OUTCOMES:
Long-term neurodevelopment: Proportion of infants who survive without neurodevelopmental disabilities at 24 months | Through study completion (average of 24 months)
Mid-term infant's general health: | Through study completion (average of 24 months)
  Proportion of infants maintaining adequate growth pattern during the first 12 months after birth
Mid-term infant's general health: | Through study completion (average of 24 months)
  proportion of infants using health system facilities after discharge
Economic impact | Through study completion (average of 24 months)
  Measure levels of resources associated with FICare implementation: The following data will be recorded:
  For neonates:
  Number of days in hospital
Economic impact | Through study completion (average of 24 months)
  Measure levels of resources associated with FICare implementation: The following data will be recorded:
  For neonates:
  Number of days on different levels of care
Economic impact | Through study completion (average of 24 months)
  Measure levels of resources associated with FICare implementation: The following data will be recorded:
  For neonates:
  Hospital readmissions (number of episodes)
Economic impact | Through study completion (average of 24 months)
  Measure levels of resources associated with FICare implementation: The following data will be recorded:
  For neonates:
  Frequentation of emergency service
Economic impact | Through study completion (average of 24 months)
  Measure levels of resources associated with FICare implementation: The following data will be recorded:
  For carers :
  Number of siblings on care
Economic impact | Through study completion (average of 24 months)
  Measure levels of resources associated with FICare implementation: The following data will be recorded for carers :
  Relation to the newborn on care: parent, legal tutor, other family member
Economic impact | Through study completion (average of 24 months)
  Measure levels of resources associated with FICare implementation: The following data will be recorded for carers :
  average hours/day on care
Economic impact | Through study completion (average of 24 months)
  Measure levels of resources associated with FICare implementation: The following data will be recorded for carers :
  overnight stay at hospital/nearby: number of overnight stays
Economic impact | Through study completion (average of 24 months)
  Measure levels of resources associated with FICare implementation: The following data will be recorded for carers :
  Payment for overnight stay
Economic impact | Through study completion (average of 24 months)
  Measure levels of resources associated with FICare implementation: The following data will be recorded for carers :
  travel to hospital for care: expenses/travel, N of trips
Economic impact | Through study completion (average of 24 months)
  Measure levels of resources associated with FICare implementation: The following data will be recorded for carers :
  other dependents under your care: N of dependents
Economic impact | Through study completion (average of 24 months)
  Measure levels of resources associated with FICare implementation: The following data will be recorded for carers :
  helps received for dependents
Economic impact | Through study completion (average of 24 months)
  cost-effectiveness estimates compareing current care to previous care model.
  The cost-effectiveness analysis of the FICare implementation will be carried out using a decision-analytical model that will be developed and populated with costs and effectiveness data from the pilot studies. For each FICare implementation site the cost-effectiveness of the intervention will be estimated as follows:
  ICER= ∆C/∆E where: ICER - incremental cost-effectiveness ratio.
  * C - difference in mean costs for post- and pre-intervention.
  * E - difference in mean effectiveness outcomes for post-and pre-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Adelina Pellicer, MD, Principal Investigator — Hospital Universitario La Paz
Locations (2):
- Hospital Universitario La Paz, Madrid, Spain
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alferink MT, Moreno-Sanz B, Cabrera-Lafuente M, Ergenekon E, de Haan TR, van Kempen AAMW, Lakhwani J, Rabe H, Zaharie GC, Pellicer A; RISEinFAMILY Consortium (European Union, MSCA-RISE-H2020). RISEinFAMILY project: the integration of families at neonatal intensive care units (NICUs) to empower them as primary caregivers: study protocol for a stepped wedge cluster controlled trial. Trials. 2024 Apr 10;25(1):248. doi: 10.1186/s13063-024-08043-7. PMID 38594733